CLINICAL TRIAL: NCT03256149
Title: Effect of High Dose Steroids on Dysphagia After Anterior Spinal Surgery: a Randomized Controlled Trial
Brief Title: High Dose Steroids for Dysphagia
Acronym: SHDD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough patients recruted
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: CE 14.247
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Dysphagia; Cervical Spine Disease
MeSH Terms: conditions — Deglutition Disorders | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Dexamethasone, 4 mg IV given at 8 hours interval, first dose received at the time of surgery (induction), 3 doses total
  Interventions: Drug: Dexamethasone
- Placebo group (Placebo Comparator): Saline given at 8 hours interval, first dose received at the time of surgery (induction), 3 doses total
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone
  Other Names: Decradron
  Arms: Treatment group
Drug: Placebo — Normal saline (IV placebo)
  Other Names: Saline
  Arms: Placebo group

SUMMARY:
Few existing data currently indicates that anti-inflammatory drugs could help diminish the local cervical inflammation tough to cause the dysphagia, hoarseness and dyspnea after an anterior surgical approach to the spine. This study aims to evaluate the effect of high dose of steroids on dysphagia after an anterior cervical spine procedure. Patients subjected to a cervical spine surgery through an anterior approach will be randomized to a treatment group receiving 3 doses of IV dexamethasone (decadron) and a placebo group receiving saline. Outcome will be measured with dysphagia scales, modified barium swallow and rhino-pharyngo-laryngoscopy, all done pre and post-operatively. Secondary outcomes involve neurological condition, pain and fusion rate.

ELIGIBILITY:
Inclusion Criteria:

* Anterior cervical spine surgery
* Elective surgery

Exclusion Criteria:

* Takes steroids for any reason
* Pre-existing condition leading to dysphagia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Voice evaluation | First day post-operatively
  Voice handicap index
Dysphagia evaluation: MBSimp | First day post-operatively
  Modified Barium Swallow with the calculation fof the MBSimp score
Soft tissue edema | First day post-operatively
  Pre-vertebral soft tissue edema on X Ray
Airway evaluation | First day post-operatively
  Rhino-Pharyngo-Laryngoscopy
Dysphagia evaluation: Rosenbeck | First day post-operatively
  Modified Barium Swallow with calculation of the Rosenbeck score

SECONDARY OUTCOMES:
Hyperreflexia | 3 months post-operatively
  hyperreflexia assesment using osteotendinous reflexes graded on a 1 to 4 scale
Fusion rate | 6 months after surgery
  Cervical spine fusion at site of surgery seen on CT scan
Pain | 3 months after surgery
  Subjective neck pain using analog pain scale
Strenght | 3 months after surgery
  4 limbs strengh assessment on a 0 to 5 scale
Crude touch sensation | 3 months after surgery
  Presence or absence of hypoesthesia in the limbs
Surgical site infection | 3 months after surgery
  Presence or absence of superficial or deep surgical site infection

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided